CLINICAL TRIAL: NCT05879094
Title: Orthopaedic Simulation of Morton's Extension to Test the Effect on Plantar Pressures of Each Metatarsal Head in Patients Without Deformity: A Pre-post-test Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/235-E
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Healthy Subjects
Keywords: metatarsalgia; foot; orthopedics
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morton extension (Experimental): Experimental group con Morton Extension application
  Interventions: Other: Morton extension

INTERVENTIONS:
Other: Morton extension — A Morton extension with a height of 5 mm was insert from the proximal area of the first metatarsal head to the base of the proximal phalanx of the Hallux of the subjects' bare feet using a paper bandage. The material, shape, size, and thickness of the Morton Extension were the same.

SUMMARY:
The aim of this study is to simulate the orthopedic treatment called Morton's extension on non-deformed patients to check the effects on each metatarsal head on its static footprint.

DETAILED DESCRIPTION:
The objective of this study is to perform an assimilation of the orthopedic treatment called morton extension on non-deformed patients to verify the effects on each metatarsal head on its static footprint, specifically the mean pressures and before and after the application of the morton extension.

ELIGIBILITY:
Inclusion Criteria:

* no history of trauma to the foot;
* the presence of at least 10° of dorsiflexion at the ankle with the knee fully dorsiflexed;
* unrestricted motion of the functional subtalar joint of 30°;
* unrestricted motion along the longitudinal axis of the midtarsal joint of 15°;
* unrestricted nonweight-bearing motion of the first ray of at least 8 mm;
* greater than 50° of dorsiflexion of the hallux to the first metatarsal bisection during nonweight-bearing;
* age greater than 18 years and younger than 60 years;
* at the time of data collection, no lower limb dysfunction or chronic injury; and
* no evidence of a non-fixed deformity at first MTP and first metatarsal cuneiform joints.

Exclusion Criteria:

* plantar corns and calluses,
* hallux valgus and lesser toe deformities,
* diabetes,
* any abnormality in the lower extremity that may affect gait.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Before Morton Extension Medium pressure | Through study completion, an average of 1 week
  Static footprint will measure medium plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
Before Morton Extension Maximum pressure | Through study completion, an average of 1 week
  Static footprint will measure maximum plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
After Morton Extension Medium pressure | Through study completion, an average of 1 week
  Static footprint will measure medium plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.
After Morton Extension Maximum pressure | Through study completion, an average of 1 week
  Static footprint will measure maximum plantar pressures of first, second third fourth fifth and midfoot rearfoot and forefoot in Kilopascals (KPa). Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline.

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Martínez-Jimenez, PhD, Principal Investigator — Mayuben Private Clinic
Locations (1):
- Eva María Martínez-Jimenez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Serena A, Losa-Iglesias ME, Becerro-de-Bengoa-Vallejo R, Morales-Ponce A, Soriano-Medrano A, Perez-Boal E, Grande-Del-Arco J, Casado-Hernandez I, Martinez-Jimenez EM. Orthopaedic Simulation of a Morton's Extension to Test the Effect on Plantar Pressures of Each Metatarsal Head in Patients without Deformity: A Pre-Post-Test Study. Diagnostics (Basel). 2023 Sep 28;13(19):3087. doi: 10.3390/diagnostics13193087. PMID 37835830